CLINICAL TRIAL: NCT06018038
Title: A Comparison of Upper Extremity Exercise Capacity, Maximum Oxygen Consumption, Daily Activities, and Physical Activity Level in Breast Cancer and Healthy Individuals
Brief Title: Arm Exercise Capacity and Maximal Oxygen Consumption With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Associate Professor, Hacettepe University
Other Study IDs: GO 23/489
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Upper Extremity; Oxygen Consumption; Healthy
Keywords: Maximal Oxygen Consumption; breast cancer; Upper Extremity Exercise Capacity; Physical Activity Level
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Breast Cancer Group: Inclusion criteria were to be between 18-65 years of age, to volunteer to participate in the study, to have Stage I-III breast cancer, to have at least 15 months after breast cancer surgery, to have six months after active breast cancer treatment (i.e. surgery/chemotherapy), to have no problems in reading and/or understanding the scales and to be able to cooperate with the tests. Exclusion criteria were the presence of active infection, musculoskeletal and neurologic disease that may affect exercise performance, symptomatic heart disease, neurologic disease or other clinical diagnosis that may affect cognitive status.
  Interventions: Diagnostic Test: Maximal Exercise Capacity, Maximal Oxygen Consumption (VO2max)
- Control Group: The inclusion criteria were to be between 18-65 years of age, to be willing to participate in the study, to have no problems in reading and/or understanding the scales and to be able to cooperate with the tests. Exclusion criteria were having any orthopedic or neuromuscular condition that would interfere with walking or exercise performance, having any chronic disease, or having psychiatric disorders or mental disorders that might interfere with cooperation or compliance with exercise tests.
  Interventions: Diagnostic Test: Maximal Exercise Capacity, Maximal Oxygen Consumption (VO2max)

INTERVENTIONS:
Diagnostic Test: Maximal Exercise Capacity, Maximal Oxygen Consumption (VO2max) — Cardiopulmonary Exercise Testing (CPET)

SUMMARY:
Breast cancer is the most common type of cancer among women worldwide. The incidence rate has reached approximately 16%. According to 2016 data from the Ministry of Health, the incidence of breast cancer in Turkey is 46.8 per 100,000 people and approximately 17,000 women are diagnosed with breast cancer each year. While breast cancer survival rate is 80% in developed countries, this rate varies between 40-60% in low-middle income countries. Survival can be increased with early diagnosis and more effective treatment methods. However, a wide range of treatment-related complications are observed during and/or after breast cancer treatment. Cancer survivors are exposed to a variety of direct (local/regional therapy, systemic therapy and supportive care) and indirect factors (modifiable and non-modifiable risk factors) that can have adverse effects on pulmonary, cardiovascular, hematologic and musculoskeletal components. Oxygen consumption in cancer patients may be adversely affected by aging, deconditioning, existing comorbidities, cancer pathophysiology and cancer treatments (surgery, radiation, chemotherapy and hormone therapy). Although decreased functional capacity is common after breast cancer treatment, there are few studies evaluating maximal arm exercise capacity with oxygen consumption.

DETAILED DESCRIPTION:
In recent years, thanks to the increasing treatment possibilities with the developing technology, the majority of patients show good functional recovery after breast cancer. However, it has been reported that the treatments negatively affect the functional capacity of the upper extremities, daily life, work and social activities and reduce the quality of life. It has also been reported that breast cancer-related lymphedema (BCRL) may both cause and exacerbate treatment-related complications such as decreased functional capacity of the upper extremities and worsened quality of life after breast cancer treatments. In addition, it has been found that lymphedema decreases the muscle strength and range of motion of the limb in which it develops and causes an increase in symptoms such as pain, fatigue and discomfort. These complications caused by lymphedema lead to decreased functional level of the upper extremity, activity limitations and decreased quality of life. Cardiovascular health is negatively affected after breast cancer. Decreased cardiorespiratory performance also has direct consequences on daily task performance and therefore quality of life is negatively affected.

The gold standard method of measuring cardiorespiratory exercise capacity is cardiopulmonary exercise testing (CPET). This method determines the causes of limitation during exercise and gives maximal oxygen consumption (VO2max) as a measure of maximum performance. In cancer patients, the oxygen system may be adversely affected by chemotherapy. Effects of chemotherapeutic agents on respiratory, cardiac, blood, vascular or skeletal muscle functions have been observed, potentially contributing to impaired cardiorespiratory fitness. Cardiorespiratory function is not routinely measured at any stage of breast cancer treatment and CPET is rarely used in clinical settings. Although low VO2max measurements have been observed in intervention studies during breast cancer survivorship and these studies were conducted without the use of an arm ergometer, to our knowledge, there is very limited information on the impact of cancer treatment on cardiorespiratory fitness using gold standard testing methods.

Although decreased functional capacity is common after breast cancer treatment, there are few studies evaluating maximal arm exercise capacity with oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

Breast Cancer Group:

1. Being between 18-65 years of age,
2. Volunteering to participate in the research,
3. Stage I-III breast cancer,
4. At least 15 months after breast cancer surgery,
5. Six months after active breast cancer treatment (i.e. surgery/chemotherapy),
6. No lymphedema
7. No problems in reading and/or understanding the scales and being able to cooperate with the tests,

Healthy group:

1. Age between 18-65 years,
2. Volunteering to participate in the research,
3. No problems in reading and/or understanding the scales and being able to cooperate with the tests.

Exclusion Criteria:

Breast Cancer Group:

1. Presence of active infection,
2. Musculoskeletal and neurological diseases that may affect exercise performance, symptomatic heart disease,
3. Having a neurological disease or other clinical diagnosis that may affect cognitive status.

Healthy group:

1. Having any orthopedic or neuromuscular condition that would interfere with walking or exercise performance,
2. Having any chronic disease or psychiatric disorders or mental impairments that may interfere with cooperation or compliance with exercise tests

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients between the ages of 18-65 years who are diagnosed with breast cancer at Hacettepe University Hospital, Department of Internal Medicine, Division of Medical Oncology, and who volunteer to participate in the study will be included in the study. For healthy groups, age and gender appropriate volunteers will be recruited for the study
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Testing (CPET) | One Year
  Maximal Oxygen Consumption (VO2max)

SECONDARY OUTCOMES:
Upper Extremity Oxidative Muscle Metabolism | One Year
  Muscle Oxygen Saturation (SmO2 )
Peripheral Muscle Strength | One Year
  Hand grip strength by hand dynamometer
Evaluation of Quality of Life | One Year
  European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) All scores were linearly transformed to a 0 to 100 scale. A high or healthy level of functioning is represented by a high functional score
Physical activity levels | One Year
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) The physical activity status of participants was grouped as follows: (a) inactive [≤600 metabolic equivalent MET)-min/week]; (b) minimum active (>600 up to ≤3000 MET-min/week); and (c) active (>3000 MET-min/week)
Upper Limb Functionality | One Year
  Upper Limb Functional Test (ULIFT)
Pain Assessment | One Year
  McGill Pain Scale McGill pain scale determines the severity of pain and is divided into zero, which means no pain, and 10, which means severe pain;
Fatigue Measurement | One Year
  Piper Fatigue Scale (PFS) Responses for each item It is evaluated between 0-10 points. The total fatigue score is based on 22 items scores are summed and divided by the number of items. Scale obtained from high scores indicate a high level of perceived fatigue shows.
anthropometric measurements | One Year
  Arm Circumference

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Principal Investigator — Hacettepe University; Melda Saglam, PhD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No